CLINICAL TRIAL: NCT06130150
Title: Evaluation of Sexual Function in High-risk Pregnant Women
Brief Title: Sexual Function in High-risk Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Cagdas Nurettin Emeklioglu, MD, Karabuk University
Other Study IDs: KBU-EMEKLIOGLU-002
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: High Risk Pregnancy; Sexual Dysfunction; Anxiety; Female Sexual Function
Keywords: high-risk pregnancy; perinatology; sexual dysfunction; female sexual function; fsfi
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk: This group includes pregnant women with the risk factors determined in the study
- Normal: This group includes pregnant women with no risk

SUMMARY:
Our aim with this study is to evaluate the sexual functions of pregnant women whose pregnancies are defined as high-risk pregnancies and whose pregnancies are followed by perinatology specialists.

ELIGIBILITY:
Inclusion Criteria: - Pregnant women over 18 years old, -Pregnant women 39 years old and under, -Pregnant women in their 3rd trimester.

Exclusion Criteria: - Pregnant women under 18 years old, -Pregnant women over 40 years old, -Pregnant women in their 1st or 2nd trimester.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women between the ages of 18-40 who were diagnosed with risky pregnancy for any reason during their pregnancy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
1 | 1 day
  High-risk pregnant women have lower FSFI score results then normal pregnant women

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Sisli, Turkey (Türkiye)